CLINICAL TRIAL: NCT07219745
Title: Transanal Irrigation for the Management of Early Low Anterior Resection Syndrome (LARS): A Pilot Randomized Controlled Trial
Brief Title: Transanal Irrigation for the Management of Early Low Anterior Resection Syndrome (LARS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE3225
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer; Low Anterior Resection Syndrome
Keywords: Transanal irrigation; Peristeen Transanal Irrigation System; Low Anterior Resection Syndrome; LARS
MeSH Terms: conditions — Colorectal Neoplasms; Low Anterior Resection Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Transanal Irrigation (TAI) - intervention arm (Other): Participants in the TAI-intervention arm will receive TAI (using Peristeen Plus Irrigation kit), training of TAI administration, and access to the LARS app (including TAI module).
  Interventions: Device: Peristeen Plus Irrigation kit; Other: LARS mobile application
- Continued conservative management - control arm. (Other): Participants in the control arm will receive conservative management and access to the LARS app (excluding the TAI module). Conservative management includes individualized combinations of dietary modifications, pharmacologic therapies, pelvic floor rehabilitation, and structured follow-up
  Interventions: Other: LARS mobile application

INTERVENTIONS:
Device: Peristeen Plus Irrigation kit — Transanal irrigation TAI is performed by inserting an applicator into the anal canal, inflating a balloon to occlude passage of stool and then installing 500-1000 mL of tap water via an irrigation system to fill the rectum and distal colon, followed by evacuation of bowel contents.
  Participants in the TAI-intervention arm will receive in-person training to learn how to use TAI and will also be given weekly virtual or in-person follow-up appointments for the first 4 weeks to troubleshoot any issues with TAI.
  Participants will do TAI once per day for 3 months. Each session of TAI takes about 20-60 minutes, depending on the individual's experience and bowel response.
  Arms: Transanal Irrigation (TAI) - intervention arm
Other: LARS mobile application — Both arms will receive access to the LARS mobile application, which is a digital self-management tool. The app provides interactive educational content, personalized bowel function diaries, guided video tutorials, and peer testimonials, all designed to enhance engagement, promote self-efficacy, and support long-term self-management.
  The TAI-intervention arm will also receive access to a TAI Module on the LARS app that will offer comprehensive educational resources, including step-by-step guidance, animations, photographs, and participant videos to reinforce safe and confident use of the TAI system.

SUMMARY:
Transanal irrigation (TAI) has shown to improve fecal incontinence and increase quality of life in patients with low anterior resection syndrome (LARS). This trial is a small study being conducted to determine whether a larger trial is feasible. Investigators are also doing this research to see if TAI impacts quality of life and improves bowel function within the early post-operative period (1-12 months).

This treatment is designed for participants to have more control over their bowel movements and reduce the dependency on immediate access to the toilet.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer in the U.S. with 152,810 new cases estimated for 2024. Rectal cancer comprises one-third of all incident cases, with rising incidence among young individuals (1-2% rise/year). With advances in multidisciplinary management, the overall, 5-year survival has improved (68%), and for localized rectal cancers it is excellent (90%), creating a growing rectal cancer survivorship population (currently >450,000). Traditionally, surgery for rectal cancer required removal of the rectum and the anus, with the creation of a permanent ostomy. However, with recent advances in subspecialty training and technique, in combination with neoadjuvant radiation, surgeons can offer a cure while preserving the anal sphincter and restoring bowel continuity, via a newer technique called Low Anterior Resection (LAR). This technique, favored by surgeons and patients, aims to allow patients to have an option of remaining "close to normal", as opposed to having a permanent ostomy. While this technique has been successful in sparing the rectum, these advancements have not come without consequence. Bowel dysfunction post-LAR, known as Low Anterior Resection Syndrome (LARS), is perhaps the most prevalent and significant sequela, affecting up to 70-90% of rectal cancer survivors. LARS symptoms include fecal incontinence, urgency, increased frequency, stool fragmentation, and incomplete evacuation. These uncontrolled LARS symptoms have a devastating impact on patients' quality of life (QoL), and often persist indefinitely. Treatment for LARS focuses on symptom management, using diet, medications and pelvic floor physiotherapy, but these measures often fail leaving patients with significant symptoms. Consequently, many patients are unable to return to work in their prior roles and require long-term disability or early retirement. Patients also resort to lifestyle restrictions including skipping meals, restricting social and recreational activities, and avoiding travel and exercise, thereby further diminishing their QoL .

Transanal irrigation (TAI) is an established treatment used for fecal incontinence and constipation. TAI is designed to irrigate a large amount of water throughout the entire colon, allowing for scheduled and complete emptying of stool. As such, TAI has the potential to reduce the symptoms of LARS including difficulty emptying, incontinence, and frequent, unpredictable bowel movements. This single daily irrigation is designed to allow patients to be free of bowel movements during the day and reduce their dependency on immediate access to the toilet, thus decreasing the impact of LARS on their daily lives. Currently, TAI is not in wide clinical use for LARS in North America despite reports from small prospective European studies (15-37 patients) demonstrating benefits for LARS . The most recent and robust published study to date, included patients with late LARS (>1-year post-treatment) randomized to TAI (n=16) vs. control (n=22), and reported significant improvements in LARS and QoL at 1 year when using TAI.

Prior work: Investigators have conducted a multi-center, cross-over, pragmatic randomized controlled trial (RCT) to assess TAI for late LARS (median 2 years post-treatment) at 7 Canadian institutions (NCT04469426). The trial has completed accrual (n=71). Patients were randomized (1:1 ratio) to start in either the TAI or control group, and then crossed over to the opposite group. Participants spent 3 months in each arm. Participants in the TAI arm received nursing instruction and online education for learning TAI using the "LARS-TAI" app. I created this web-based HIPAA-compliant, mobile app (iOS™ and Android™ compatible) to support patients with LARS using TAI. The LARS-TAI App is accessible on any device with internet access or cellular data, including smart phones, tablets, and computers. The app contains educational modules on LARS and TAI, a discussion forum, patient videos, and bowel diaries. Investigators are currently completing follow-up and data analysis for this study. This cross-over trial has provided invaluable practical knowledge on educating patients about TAI and has demonstrated a high level of acceptance for TAI as a treatment for LARS within the first North American sample. Furthermore, it has underscored the challenges associated with a cross-over study design, as many participants were hesitant to transition from TAI to the control group due to the marked improvements in LARS and QoL that they experienced with the intervention.

At CCF-FL, I have established a LARS Clinic, with a trained LARS nurse, and investigators have treated over 50 rectal cancer patients with LARS in 2024. Investigators have established a LARS registry and are routinely screening for LARS in our rectal cancer patients. Investigators have partnered with CCF-Ohio who have also started screening rectal cancer patients for LARS. Investigators have identified a high burden (75% major LARS) of LARS post-treatment in our rectal cancer patients.

The knowledge gap: While TAI shows promise for LARS management, the optimal timing for its use remains unclear. The first 6 months post-treatment pose significant challenges for LARS patients, with at least 58% experiencing major LARS and significantly decreased quality of life (QoL). Investigators observed that 54% of these patients with major LARS also experience financial distress, with most unable to return to work. Unfortunately, conservative measures often fail in this early phase, rendering patients in despair as they try to adapt to their altered bowel function. The potential for TAI to improve LARS in this early phase was proposed in a small German RCT (n=37) that demonstrated reduced bowel movements and improved LARS with no significant complications .

Overall, TAI has only been reported in 9 published studies (total n=204) all from outside of the US, including only 3 small RCTs (total n=102). Although these trials are somewhat limited in size and design, taken together they represent important evidence for the benefit of TAI in LARS and are the basis for pursuing a larger North American RCT. TAI is promising for decreasing LARS and improving QoL. Despite this available evidence on the potential benefits of TAI for LARS, TAI is currently not in standard clinical use for LARS in North America due to limited North American data. As such, TAI for the indication of LARS is not available to patients and current insurance plans (medicare/medicaid or private) do not cover its cost. This pilot trial aims to assess the feasibility of a larger trial that will build on the foundation of evidence that supports the use of TAI in rectal cancer patients with LARS. In this pilot and subsequent larger trial, investigators will gather North American data to support the use of TAI in a North American population, especially in the early post-treatment period.

Expected Results: Investigators hypothesize that TAI will decrease early LARS and positively impact quality of life for rectal cancer patients. Investigators aim to transition into a phase III study, with pilot study cases contributing to the larger sample. This strategy optimizes pilot study data use, maintains research momentum, and builds on initial findings. Successful pilot completion will yield data affirming TAI's feasibility and potential efficacy in managing LARS, bolstering our applications for extramural funding (NIH R01 Research Project Grant).

Impact: More than 450,000 rectal cancer patients in the US will enter survivorship for rectal cancer this year, with a rising number of younger patients of working age affected by rectal cancer. TAI may help patients significantly control their symptoms from the early post-operative period, allowing them to return to work and normal activities sooner and improve their QoL. The success of this pilot and consequently our larger trial will provide the necessary evidence to incorporate TAI into standard practice for LARS treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years-old) patients who underwent a LAR for any indication via open, laparoscopic, robotic, or transanal total mesorectal excision, with creation of a diverting loop ileostomy,
2. have confirmed anastomotic healing demonstrated by flexible sigmoidoscopy and CT scan with rectally-administered water soluble contrast or gastrograffin enema,
3. are planned for an ileostomy closure operation, and
4. are in the first 12 months post-LAR operation

Exclusion Criteria:

1. Inability to comprehend English or Spanish or provide informed consent (Note: after the English documents are approved, the study team plans to obtain a Spanish consent and study documents),
2. ongoing chemotherapy or radiotherapy, and
3. ongoing anastomotic complication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS)-GI Diarrhea at baseline | Baseline
  PROMIS_GI Diarrhea with domains covering Frequency, urgency, burden. T-score (mean = 50, SD = 10); higher scores = worse diarrhea
Patient-Reported Outcomes Measurement Information System (PROMIS)-GI Diarrhea at 1 month | 1 month post randomization
  PROMIS_GI Diarrhea with domains covering Frequency, urgency, burden. T-score (mean = 50, SD = 10); higher scores = worse diarrhea
Patient-Reported Outcomes Measurement Information System (PROMIS)-GI Diarrhea at 2 months | 2 months post randomization
  PROMIS_GI Diarrhea with domains covering Frequency, urgency, burden. T-score (mean = 50, SD = 10); higher scores = worse diarrhea
Patient-Reported Outcomes Measurement Information System (PROMIS)-GI Diarrhea at 3 months | 3 months post randomization
  PROMIS_GI Diarrhea with domains covering Frequency, urgency, burden. T-score (mean = 50, SD = 10); higher scores = worse diarrhea
PROMIS-GI Fecal Incontinence at baseline | Baseline
  PROMIS_GI Fecal Incontinence with domains covering Leakage, control, impact . T-score (mean = 50, SD = 10); higher scores = worse incontinence
PROMIS-GI Fecal Incontinence at 1 month | 1 month post randomization
  PROMIS_GI Fecal Incontinence with domains covering Leakage, control, impact . T-score (mean = 50, SD = 10); higher scores = worse incontinence
PROMIS-GI Fecal Incontinence at 2 months | 2 months post randomization
  PROMIS_GI Fecal Incontinence with domains covering Leakage, control, impact . T-score (mean = 50, SD = 10); higher scores = worse incontinence
PROMIS-GI Fecal Incontinence at 3 months | 3 months post randomization
  PROMIS_GI Fecal Incontinence with domains covering Leakage, control, impact . T-score (mean = 50, SD = 10); higher scores = worse incontinence
Average monthly randomization rate | 3 months post ileostomy
  Participants who report a LARS Score of ≥20-the threshold for moderate-to-severe LARS-will meet criteria for randomization. Score range: 0-42 (higher scores = more severe LARS; 0-20 = no LARS, 21-29 = minor, 30-42 = major)

SECONDARY OUTCOMES:
PROMIS Physical Function at baseline | Baseline
  PROMIS_Physical Function with domains covering Physical capability, daily activity performance.T-score (mean = 50, SD = 10); higher scores = better physical function
PROMIS Physical Function at 1 month | 1 month post randomization
  PROMIS_Physical Function with domains covering Physical capability, daily activity performance.T-score (mean = 50, SD = 10); higher scores = better physical function
PROMIS Physical Function at 2 months | 2 months post randomization
  PROMIS_Physical Function with domains covering Physical capability, daily activity performance. T-score (mean = 50, SD = 10); higher scores = better physical function
PROMIS Physical Function at 3 months | 3 months post randomization
  PROMIS_Physical Function with domains covering Physical capability, daily activity performance.T-score (mean = 50, SD = 10); higher scores = better physical function
PROMIS Ability to Participate in Social Roles and Activities at baseline | Baseline
  PROMIS_Ability to Participate in Social Roles and Activities with domains covering Social, role functioning, engagement in daily life. T-score (mean = 50, SD = 10); higher scores = better social participation
PROMIS Ability to Participate in Social Roles and Activities at 1 month | 1 month post randomization
  PROMIS_Ability to Participate in Social Roles and Activities with domains covering Social, role functioning, engagement in daily life. T-score (mean = 50, SD = 10); higher scores = better social participation
PROMIS Ability to Participate in Social Roles and Activities at 2 months | 2 months post randomization
  PROMIS_Ability to Participate in Social Roles and Activities with domains covering Social, role functioning, engagement in daily life. T-score (mean = 50, SD = 10); higher scores = better social participation
PROMIS Ability to Participate in Social Roles and Activities at 3 months | 3 months post randomization
  PROMIS_Ability to Participate in Social Roles and Activities with domains covering Social, role functioning, engagement in daily life. T-score (mean = 50, SD = 10); higher scores = better social participation
PROMIS Anxiety at baseline | Baseline
  PROMIS_anxiety with domains covering Anxiety symptoms. T-score (mean = 50, SD = 10); higher scores = more anxiety
PROMIS Anxiety at 1 month | 1 month post randomization
  PROMIS_anxiety with domains covering Anxiety symptoms. T-score (mean = 50, SD = 10); higher scores = more anxiety
PROMIS Anxiety at 2 months | 2 months post randomization
  PROMIS_anxiety with domains covering Anxiety symptoms. T-score (mean = 50, SD = 10); higher scores = more anxiety
PROMIS Anxiety at 3 months | 3 months post randomization
  PROMIS anxiety with domains covering Anxiety symptoms. T-score (mean = 50, SD = 10); higher scores = more anxiety
PROMIS Depression at baseline | Baseline
  PROMIS depression with domains covering Depressive symptoms .T-score (mean = 50, SD = 10); higher scores = more depression
PROMIS Depression at 1 month | 1 month post randomization
  PROMIS depression with domains covering Depressive symptoms .T-score (mean = 50, SD = 10); higher scores = more depression
PROMIS Depression at 2 months | 2 months post randomization
  PROMIS depression with domains covering Depressive symptoms .T-score (mean = 50, SD = 10); higher scores = more depression
PROMIS Depression at 3 months | 3 months post randomization
  PROMIS depression with domains covering Depressive symptoms .T-score (mean = 50, SD = 10); higher scores = more depression
PROMIS Sleep Disturbance at baseline | Baseline
  PROMIS Sleep Disturbance with domains covering Sleep quality, falling/ staying asleep, restfulness. T-score (mean = 50, SD = 10); higher scores = more sleep disturbance
PROMIS Sleep Disturbance at 1 month | 1 month post randomization
  PROMIS Sleep Disturbance with domains covering Sleep quality, falling/ staying asleep, restfulness. T-score (mean = 50, SD = 10); higher scores = more sleep disturbance
PROMIS Sleep Disturbance at 2 months | 2 months post randomization
  PROMIS Sleep Disturbance with domains covering Sleep quality, falling/ staying asleep, restfulness. T-score (mean = 50, SD = 10); higher scores = more sleep disturbance
PROMIS Sleep Disturbance at 3 months | 3 months post randomization
  PROMIS Sleep Disturbance with domains covering Sleep quality, falling/ staying asleep, restfulness. T-score (mean = 50, SD = 10); higher scores = more sleep disturbance
PROMIS Satisfaction with Social Roles at baseline | Baseline
  PROMIS Satisfaction with Social Roles, with domains covering Satisfaction with role & social engagement. T-score (mean = 50, SD = 10); higher scores = greater satisfaction
PROMIS Satisfaction with Social Roles at 1 month | 1 month post randomization
  PROMIS Satisfaction with Social Roles, with domains covering Satisfaction with role & social engagement. T-score (mean = 50, SD = 10); higher scores = greater satisfaction
PROMIS Satisfaction with Social Roles at 2 months | 2 months post randomization
  PROMIS Satisfaction with Social Roles, with domains covering Satisfaction with role & social engagement. T-score (mean = 50, SD = 10); higher scores = greater satisfaction
PROMIS Satisfaction with Social Roles at 3 months | 3 months post randomization
  PROMIS Satisfaction with Social Roles, with domains covering Satisfaction with role & social engagement. T-score (mean = 50, SD = 10); higher scores = greater satisfaction
PROMIS Self-Efficacy for Managing Chronic Conditions at baseline | Baseline
  PROMIS Self-Efficacy for Managing Chronic Conditions, with domains covering Satisfaction with Confidence in managing symptoms and health tasks. T-score (mean = 50, SD = 10); higher scores = greater self-efficacy
PROMIS Self-Efficacy for Managing Chronic Conditions at 1 month | 1 month post randomization
  PROMIS Self-Efficacy for Managing Chronic Conditions, with domains covering Satisfaction with Confidence in managing symptoms and health tasks. T-score (mean = 50, SD = 10); higher scores = greater self-efficacy
PROMIS Self-Efficacy for Managing Chronic Conditions at 2 months | 2 months post randomization
  PROMIS Self-Efficacy for Managing Chronic Conditions, with domains covering Satisfaction with Confidence in managing symptoms and health tasks. T-score (mean = 50, SD = 10); higher scores = greater self-efficacy
PROMIS Self-Efficacy for Managing Chronic Conditions at 3 months | 3 months post randomization
  PROMIS Self-Efficacy for Managing Chronic Conditions, with domains covering Satisfaction with Confidence in managing symptoms and health tasks. T-score (mean = 50, SD = 10); higher scores = greater self-efficacy
Completeness | 3 months post randomization
  Proportion of participants completing the 3-month outcome assessment.
Treatment adherence rate | 3 months post randomization
  Proportion of participants completing at least 80% of TAI sessions over 3-months
Consent rates | Post consenting, Baseline
  Proportion of participants undergoing ileostomy closure who provide informed consent.

CONTACTS AND LOCATIONS:
Locations (1):
- Case Comprehensive Cancer Center, Digestive Disease Institute Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: The data will be kept in a de-identified manner for 10 years following study completion. The data will then be reported anonymously and kept indefinitely.